CLINICAL TRIAL: NCT00941577
Title: A Phase 2a, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Bronchial Allergen Challenge Study to Assess the Safety, Tolerability, and Efficacy of Inhaled AIR645 in Subjects With Mild Allergic Asthma
Brief Title: Study Evaluating the Effects of AIR645 on Allergen-Induced Airway Responses in Subjects With Mild Atopic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altair Therapeutics, Inc. (Industry)
Responsible Party: Mike Hodges, MD - Chief Medical Officer, Altair Therapeutics Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIR645-CS2
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Asthma
Keywords: Hypersensitivity; Lung Diseases, Obstructive; Immune System Diseases; Respiratory Tract Diseases; Bronchial Diseases; Lung Diseases; Hypersensitivity, Immediate; Asthma; Respiratory Hypersensitivity
MeSH Terms: conditions — Asthma; Hypersensitivity; Lung Diseases, Obstructive; Immune System Diseases; Respiratory Tract Diseases; Bronchial Diseases; Lung Diseases; Hypersensitivity, Immediate; Respiratory Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR645 (Experimental): AIR645 (an IL-4/IL-13 dual cytokine signaling inhibitor) solution (diluent: physiologic saline solution)
  Interventions: Drug: AIR645
- Physiologic saline solution (Placebo Comparator): Physiologic saline solution
  Interventions: Drug: Physiologic saline solution

INTERVENTIONS:
Drug: AIR645 — AIR645 (blinded) by nebulization, range of doses, maximum of one dose per day, maximum of 6 doses in 22 days.
  Arms: AIR645
Drug: Physiologic saline solution — Placebo (blinded) by nebulization, range of doses, maximum of one dose per day, maximum of 6 doses in 22 days.
  Arms: Physiologic saline solution

SUMMARY:
To assess the efficacy of inhaled AIR645 in the suppression of the Asthmatic Responses in subjects with mild asthma inhaling an allergen.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with well controlled mild allergic asthma, aged 18 to 65 years
* Only asthma med is short-acting bronchodilator used not more than twice weekly
* FEV1 greater than 70% predicted and a demonstrated baseline late response to allergen induction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the percentage decrease forced expiratory volume in one second (FEV1) from baseline between AIR645 and placebo | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Mike Hodges, MD, Study Director — Altair Therapeutics, Inc.
Locations (3):
- Canada (3):
  - Hamilton, Ontario
  - Laval, Quebec
  - Saskatoon, Saskatchewan